CLINICAL TRIAL: NCT02267408
Title: A Single-site, Randomized Controlled Feasibility Trial of the Fearon Algorithm to Improve Management of Patients With Unstable Warfarin Effect.
Brief Title: Randomized Controlled Feasibility Trial of the Fearon Algorithm to Improve Management of Unstable Warfarin
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated by sponsor
Sponsor: McMaster University (Other)
Collaborators: Epitome Pharmaceuticals (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fearon pilot RCT, version 03
Record Dates: First submitted 2014-10-14; First posted 2014-10-17 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2016-03

CONDITIONS: Hypoprothrombinemia
Keywords: Heart valve prosthesis; Anticoagulation; Warfarin
MeSH Terms: conditions — Hypoprothrombinemias

STUDY DESIGN:
Intervention Model Description: Dosing of warfarin according to the Fearon algorithm or routine during 6 months for patients with unstable INRs
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fearon algorithm dosing (Experimental): Warfarin adjustment using the Fearon algorithm
  Interventions: Other: Warfarin adjustment using the Fearon algorithm
- Standard dosing (Active Comparator): Warfarin adjustment using standard dosing
  Interventions: Other: Warfarin adjustment using standard dosing

INTERVENTIONS:
Other: Warfarin adjustment using the Fearon algorithm — All available historical data will be used to calculate with the Fearon algorithm the individual sensitivity to warfarin and to dose changes as well as lag time until a dose adjustment reaches full effect. Based on this a personal dosing nomogram will be developed and provided to the investigator and to the patients. This nomogram will be used during 6 month but override is possible if the investigator feels that the suggestion from the nomogram is unsafe.
  Arms: Fearon algorithm dosing
Other: Warfarin adjustment using standard dosing — Patients will receive warfarin dosing instructions from a trained nurse using fixed nomograms and computer-based dosing suggestion.
  Arms: Standard dosing

SUMMARY:
Patients on warfarin but with unstable international normalized ratio (INR) will be recruited to a randomized trial comparing dosing based on an algorithm (Fearon algorithm, named after the mathematician Michael Fearon), which uses historical data to estimate patients' sensitivity to warfarin and to dose changes as well as the lag time until a dose adjustment takes effect, or to the investigators standard management Main outcome is improvement in time in therapeutic range.

DETAILED DESCRIPTION:
Patients with very variable INRs resulting in a low proportion of time in therapeutic range (TTR) have a higher risk of both bleeding complications and thromboembolic events. A good TTR is generally considered to be over 60% and "excellent TTR" is above 72% of time in range. The investigators will recruit patients with a TTR below 50%.

The Fearon algorithm provides a more thorough understanding of the individual responses to changes in warfarin dose and with a personalized nomogram for dose adjustments and timing of laboratory tests the investigators have an opportunity to improve the TTR and on a larger scale to reduce clinically important adverse events. Before embarking on a large randomized trial with this revised Fearon algorithm-derived nomogram this pilot study with a randomized, open-label design will be performed to demonstrate proof of principle.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mechanical heart valve prosthesis managed for the warfarin therapy by the Thrombosis Service at HHS-General Hospital.
* Treated with warfarin for at least 1 year.
* Therapeutic INR range 2.0-3.0 or 2.5-3.5.
* TTR in the lowest quartile

Exclusion Criteria:

* Known poor compliance due to for example alcohol abuse or cognitive impairment
* Refusal to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-11; Primary Completion 2017-02 (Actual); Study Completion 2017-02-03 (Actual)

PRIMARY OUTCOMES:
Improvement in TTR | 6 months
  The percent units of TTR during the 6 months will be compared with the percent units TTR in the previous year

SECONDARY OUTCOMES:
Proportion of patients with improvement in TTR | 6 months
  Proportion of included patients with TTR improvement of more than 5 percent units

CONTACTS AND LOCATIONS:
Overall Officials: Sam Schulman, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- Thrombosis Service, HHS-General Hospital, Hamilton, Ontario, Canada